CLINICAL TRIAL: NCT05899114
Title: Less Is More: Optimized Pharmacotherapy With Improved coNtinuity of CarE in hospitaLized oLder peOple
Acronym: LIMONCELLO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Amsterdam UMC, location AMC (Other); Amphia ziekenhuis (Unknown); Catharina Ziekenhuis Eindhoven (Other); Deventer Ziekenhuis (Other); Diakonessenhuis, Utrecht (Other); Erasmus Medical Center (Other); HagaZiekenhuis (Other); Leiden University Medical Center (Other); Meander Medisch Centrum (Other); University Medical Center Groningen (Other); UMC Utrecht (Other); Zaans Medisch Centrum (Other); Ziekenhuisgroep Twente (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Zorgevaluatie Nederland (Unknown); Canisius Wilhelmina Ziekenhuis (CWZ) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NL82393.091.22; 10330032010002 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2023-05-23; First posted 2023-06-12 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Polypharmacy; Medication Review
Keywords: Polypharmacy; Medication Review; Aged; Deprescribing

STUDY DESIGN:
Intervention Model Description: Cluster randomized study
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor, assessing whether a readmission is drug related will be masked.
  Masking the patients, care provider or investigator is not possible in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transitional Multidisciplinary Pharmacotherapeutic Care (TMPC) (Experimental): The participants in hospitals allocated to the intervention arm will receive TMPC, which will be executed by a Pharmacotherapy-team and will take place during the index hospital stay. This Pharmacotherapy-team will be composed of a physician and a hospital pharmacist, preferably registered as clinical pharmacologists.
  Interventions: Other: Transitional Multidisciplinary Pharmacotherapeutic Care
- Usual care (No Intervention): The comparator in this study is usual care, which refers to the entire spectrum of medication-related interventions by different healthcare providers (physician, pharmacist, nurse etc.) which the patient undergoes during hospital admission.

INTERVENTIONS:
Other: Transitional Multidisciplinary Pharmacotherapeutic Care — A structured medication review with improved transitional care and multidisciplinary collaboration.
  TMPC consists of the following four elements:
  1. A structured pharmacotherapeutic analysis
  2. A transitional multidisciplinary discussion.The treating physician in the hospital will be involved. The general practitioner and community pharmacist will be consulted.
  3. An interview and discussion with the patient and/or legal representative by a member of the Pharmacotherapy-team, which will be performed before the patient is discharged from the hospital.
  4. A discharge note with the pharmacotherapeutic care plan. This will be sent to the community pharmacist and the general practitioner.
  Other Names: TMPC
  Arms: Transitional Multidisciplinary Pharmacotherapeutic Care (TMPC)

SUMMARY:
The goal of this cluster randomized controlled trial is to compare transitional multidisciplinary pharmacotherapeutic care (TMPC) with usual care in patients aged 70 years or older with polypharmacy, admitted to the hospital via the emergency department for longer than 24 hours and that have an elevated risk of drug related readmissions.

The primary aims of the study are:

* To assess whether TMPC leads to a decrease in number of DRreAs compared to usual care during the first 30 days after index hospitalisation.
* To assess whether TMPC is cost-effective

Participants will receive TMPC in hospitals allocated to the intervention. TMPC will be executed by a pharmacotherapeutic team, it consists of the following four elements:

* pharmacotherapeutic analysis
* transitional multidisciplinary discussion
* pharmacotherapeutic care interview and discussion with the patient
* discharge note with the pharmacotherapeutic care plan

Researchers will compare TMPC with usual care to assess the effect and cost-effectiveness of TMPC.

DETAILED DESCRIPTION:
Rationale: Polypharmacy poses an ongoing healthcare challenge, as it is associated with negative outcomes such as adverse drug events, lower quality of life and mortality. These risks are especially elevated for the frail and old, leading to high numbers of drug related admissions (DRAs) and unplanned emergency department visits. Approximately half of the DRAs are potentially preventable, and therefore a possible target point for interventions. Unfortunately, until now, despite multiple efforts to decrease drug related harm, the number of drug related admissions has not decreased. Several studies have previously investigated the effect of a structured medication review with varying success. Identified strengths were multicomponent approaches, multidisciplinary approaches and selection of specifically high-risk patients. The LIMONCELLO study will take this into account and will study a multidisciplinary multicomponent intervention with focus on transitional care in a patient population that is most likely to benefit from this intervention. It is hypothesised that transitional multidisciplinary pharmacotherapeutic care (TMPC) is superior in preventing drug related readmissions (DRreAs) compared to usual care.

Objective: The LIMONCELLO study aims to assess the effect and cost-effectiveness of TMPC compared to usual care.

Study design: This is a cluster randomised controlled trial, a cluster will be defined at the hospital level, with each cluster randomly allocated to the intervention or control group. Patients aged 70 years or older with polypharmacy, admitted to the hospital via the emergency department for longer than 24 hours, with completed medication verification and with an elevated risk of drug related readmissions (calculated by use of the DRA prediction model, an algorithm developed by the OPERAM study group) will be included. Participants in intervention hospitals will receive TMPC during index hospitalisation. TMPC consists of four elements: pharmacotherapeutic analysis, transitional multidisciplinary discussion, pharmacotherapeutic care interview and discussion with the patient, and a discharge note with the pharmacotherapeutic care plan. The comparator is usual care as is provided in the participating hospitals. Follow-up will be 1 year, participants will be called 30 days, 3 months and 12 months after index hospitalisation.

Statistical considerations: 16 clusters will participate in the study, requiring a total of 161 patients per cluster to be included, 2,576 participants in total. Results will be analysed by intention-to-treat analysis and per-protocol analysis. For the primary outcome, drug related readmissions, a generalized linear mixed model with a binomial distribution and logit link function will be used for the analysis on an individual level, adjusting for clustering.

ELIGIBILITY:
Inclusion Criteria:

* 70 years or older
* Polypharmacy, the use of 5 or more regular medications, defined as authorised medications with registration numbers, used for more than 30 days. Topical preparations are excluded from this definition.
* Admitted to hospital through the ED (which comprises both the general emergency department and the cardiac emergency department)
* Length of hospitalisation more than 24 hours
* Completed medication verification
* DRA prediction percentage of 23.0% or higher

Exclusion Criteria:

* No informed consent by patient or a legal representative
* Participation in an interfering clinical trial
* Elective hospital admission
* Direct admission to the ICU (when medication verification as usual can't be executed, and therefore inclusion of patients as described in 10.2 is not possible)
* A life expectancy of less than 3 months, which includes patients with palliative treatment at home, direct admission to palliative care or palliative care planned within 24 hours after index hospital admission.
* Patient or legal representative not able to speak Dutch.
* Follow-up of patient primarily by secondary caregivers. This refers to situations where the secondary caregiver is in the lead of the medication list of the patient instead of the GP or elderly care physician, for example in the following patient groups:

  * patients receiving intensive oncologic therapy
  * patients in an organ- or stem cell transplantation procedure
  * patients receiving intensive (chronic) psychiatric care, such as patients admitted to a medical psychiatric unit
  * patients on dialysis

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2576 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2026-01-17 (Estimated)

PRIMARY OUTCOMES:
Number of Drug Related Readmissions in the first 30 days after index hospitalisation | 30 days after index hospitalisation
  Whether readmission is drug related will be assessed with AT-HARM10

SECONDARY OUTCOMES:
Number of Drug Related Readmissions at 3 and 12 months after index hospitalisation | 3 and 12 months after index hospitalisation
  Whether readmission is drug related will be assessed with AT-HARM10
Duration of hospitalisation of Drug Related Readmission | 30 days, 3 months and 12 months after index hospitalisation
  Whether readmission is drug related will be assessed with AT-HARM10
Time to first Drug Related Readmission | 30 days, 3 months and 12 months after index hospitalisation
  Whether readmission is drug related will be assessed with AT-HARM10
Number of Emergency Department visits | 30 days, 3 months and 12 months after index hospitalisation
Number of all-cause hospital readmissions | 30 days, 3 months and 12 months after index hospitalisation
Healthcare costs | 30 days, 3 months and 12 months after index hospitalisation
  In euros, assessed with the iMTA Medical Consumption Questionnaire (iMCQ)
Quality of Life measured with EQ-5D-5L | 30 days, 3 months and 12 months after index hospitalisation
  Measured by 5-level EuroQol-5 domains (EQ-5D-5L) questionnaire
Cost-effectiveness | During the 12 month follow-up
  In euro per Quality Adjusted Life Year (QALY) gained, by combining costs and quality of life measurements
Number of regular medications | At discharge from index hospitalisation and 30 days, 3 months and 12 months after index hospitalisation
  Based on number of regular medications in the medication list
Number and type of recommendations in the intervention group | At discharge from index hospitalisation
  Based on documented recommendations made during TMPC
Number of implemented recommendations | 30 days, 3 months and 12 months after index hospitalisation
  The number of differences between the pharmacotherapeutic plan composed by the P-team and the participant's current medication list at each time point
Activities of Daily Living | 30 days, 3 months and 12 months after index hospitalisation
  Measured with Katz-6 ADL questionnaire
Number of patients living independently | 30 days, 3 months and 12 months after index hospitalisation
Number of falls | 30 days, 3 months and 12 months after index hospitalisation
Mortality | 30 days, 3 months and 12 months after index hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Kees Kramers, Prof. Dr., Principal Investigator — Radboud University Medical Center
Locations (16):
- Netherlands (16):
  - Canisius Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Radboudumc, Nijmegen, Gelderland
  - Amphia ziekenhuis, Breda, North Brabant
  - Catharina Ziekenhuis, Eindhoven, North Brabant
  - Amsterdam UMC - location VUMC, Amsterdam, North Holland
  - Amsterdam UMC- location AMC, Amsterdam, North Holland
  - Zaans Medisch Centrum, Zaandam, North Holland
  - Ziekenhuisgroep Twente, Almelo, Overijssel
  - Deventer Ziekenhuis, Deventer, Overijssel
  - Universitair Medisch Centrum Groningen, Groningen, Provincie Groningen
  - Leiden Universitair Medisch Centrum, Leiden, South Holland
  - Erasmus Medisch Centrum Rotterdam, Rotterdam, South Holland
  - Haga Ziekenhuis, The Hague, South Holland
  - Meander Medisch Centrum Amersfoort, Amersfoort, Utrecht
  - Diakonessenhuis, Utrecht, Utrecht
  - Universitair Medisch Centrum Utrecht, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared in a repository, published under restricted access.
Time Frame: All collected data will be stored for 15 years
Access Criteria: It will be shared in a repository. The data will be published under restricted access. Requests for access will be checked, by a data access committee (DAC) formed by the consortium.

REFERENCES:
- [Derived] Cooijmans S, Engelen EMC, Wuyts SCM, Kramers C, van Agtmael MA, van den Bemt PMLA, Bouvy ML, Amouch H, Autar RS, Benoist GE, van Berlo-van de Laar IRF, Derijks-Engwegen JYMN, van den Elsen G, Engelaer FM, Gombert-Handoko KB, Jansen DRM, Kerskes MHM, Kruik-Kolloffel WJ, Kuijvenhoven MA, van der Kuy HM, Labots G, van Poelgeest EP, Sablerolles R, Sallevelt BTG, van Stiphout F, Storm BN, Taks M, Teeuwisse PJI, Uiterwijk J, Vondeling A, de Vries M, Wesselink E, Wiggers NML, de Wit HAJM, Schers HJ, Adang EMM, van Wely M, van Herwaarden N, Knol W. Less Is More: Optimized pharmacotherapy with improved coNtinuity of CarE in hospitaLized oLder peOple (LIMONCELLO): study protocol of a cluster randomized controlled trial. BMC Geriatr. 2025 Dec 24;25(1):1034. doi: 10.1186/s12877-025-06533-0. PMID 41444867
- See also: LIMONCELLO website in collaboration with "Zorgevaluatie Nederland" — http://www.zorgevaluatienederland.nl/limoncello